CLINICAL TRIAL: NCT00495807
Title: Influence on Pain Management of Nurses' Negative Words After Total Hysterectomy
Brief Title: Nurses' Negative Words and Postoperative Pain Management
Acronym: NWPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Confidential Enquiry into Maternal and Child Health (Other)
Responsible Party: XiaoFeng Shen, Nanjing Maternal and Child Health Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NMU-2579-2FW; NMCH2006-012
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-04

CONDITIONS: Postoperative Pain
Keywords: Psychological Tests; Pain, Postoperative; Nurses
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): No Words was delivered during the PCA management
  Interventions: Behavioral: No Words
- 2 (Active Comparator): Positive words was delivered as a positive control group during the therapy of the pain with PCA
  Interventions: Behavioral: Positive words
- 3 (Active Comparator): Partially negative words was delivered during the PCA pain management
  Interventions: Behavioral: Partially Negative Words
- 4 (Active Comparator): Totally negative words was delivered during the PCA pain management
  Interventions: Behavioral: Totally Negative Words

INTERVENTIONS:
Behavioral: No Words — Without any words was given during pain management
  Other Names: NW
  Arms: 1
Behavioral: Positive words — Positive words was given to PCA pain management patients at different time point,i.e. 3h, 6h, 12h and 18h.
  Other Names: PW
  Arms: 2
Behavioral: Partially Negative Words — Partially negative words was given during PCA pain management at different time point,i.e. 3h, 6h, 12h and 18h.
  Other Names: PNW
  Arms: 3
Behavioral: Totally Negative Words — Totally negative words was given during PCA pain management at different time points, i.e. 3h, 6h, 12h and 18h
  Other Names: TNW
  Arms: 4

SUMMARY:
Psychological implications expressed pivotal effects on daily activities. Postoperative pain management is always encountered varying influence from the ambience of surgical wards, especially the nurses. We hypothesized that nurses' negative or positive words would produce unexpected role in pain management, which might be a strong factor resulting in the failure of postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Abdominal Surgery
* > 18yr < 65yr
* Female
* Administration of postoperative analgesia
* Patient-controlled analgesia

Exclusion Criteria:

* With cardiac or/and pulmonary diseases
* Allergy to Opioids
* > 20% alteration in vital signs
* Unwilling to finish the follow-up process
* Respiratory depression
* > = 65yr = < 18yr
* Non-Chinese

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale of Pain | 0h to 48h after operation

SECONDARY OUTCOMES:
Morphine consumption; VAS sedation; VAS satisfaction; Side effects; Patient's overall conditions | 0-48h after surgeries

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Wang F, Shen X, Xu S, Liu Y, Ma L, Zhao Q, Fu D, Pan Q, Feng S, Li X. Negative words on surgical wards result in therapeutic failure of patient-controlled analgesia and further release of cortisol after abdominal surgeries. Minerva Anestesiol. 2008 Jul-Aug;74(7-8):353-65. PMID 18612266